CLINICAL TRIAL: NCT01977846
Title: Natural History of Progression of Atrophy Secondary to Stargardt Disease: Retrospective, and Prospective Longitudinal Observational Study Incl. Ancillary SMART Study- Scotopic Microperimetric Assessment of Rod Function in Stargardt Disease
Brief Title: A Natural History of the Progression of Stargardt Disease: Retrospective and Prospective Studies
Acronym: ProgSTAR
Status: Completed | Type: Observational
Sponsor: Foundation Fighting Blindness (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FFBCRI-PROGSTAR-01/02
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-07

CONDITIONS: Stargardt Disease
Keywords: genetic testing; ABCA4; Stargardt; retina; retinal degeneration
MeSH Terms: conditions — Stargardt Disease; Retinal Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Stargardt disease is currently an incurable and untreatable macular dystrophy that causes severe visual loss in children and young adults, thereby causing enormous morbidity with economic, psychological, emotional, and social implications. There are no FDA approved therapeutic treatments for this disease. Therefore, the objective of this study is to collect natural history data from a large population of children and adults in order to evaluate possible efficacy measures for planned clinical trials.

Participants will be recruited from each Investigator's own patient population as the study requires the availability of both multiyear retrospective data, as well as ongoing prospectively collected data. A concurrent ancillary study (SMART study) is also being conducted with a subset of the prospective study patients during their regular ProgSTAR study visits to expand the collection of retinal images to include microperimetry measurements gathered under scotopic (low light) conditions.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed informed consent form and authorization allowing the disclosure and use of protected health information.
* The designated primary study eye must have at least one well-demarcated area of atrophy as imaged by fundus autofluorescence with a minimum diameter of 300 microns and all lesions together must add to less than or equal to 12 mm2 (equivalent to no more than 5 disc areas in a least one eye) and a BCVA of 20 ETDRS letters (20/400 Snellen equivalent) or better.
* Two (2) pathogenic mutations confirmed present, in the ABCA4 gene. If only one ABCA4 allele contains a pathogenic mutation, the patient shall have a typical Stargardt phenotype, namely at least one eye must have flecks at the level of the retinal pigment epithelium typical for STGD.
* The primary study eye must have clear ocular media and adequate pupillary dilation to permit good quality fundus autofluorescence (FAF) and Spectral-Domain optical coherence tomography (sd-OCT) imaging in the opinion of the investigator.
* Be able to cooperate in performing the examinations.
* Be willing to undergo ocular examinations once every 6 months for up to 24 months.
* Be at least six years old.
* Both eyes can be included if inclusion criteria are fulfilled for both eyes.

Exclusion Criteria:

* Ocular disease, such as choroidal neovascularization, glaucoma and diabetic retinopathy, in either eye that may confound assessment of the retina morphologically and functionally.
* Intraocular surgery in the primary study eye within 90 days prior to baseline visit.
* Current or previous participation in an interventional study to treat STGD such as gene therapy or stem cell therapy. Current participation in a drug trial or previous participation in a drug trial within six months before enrollment. The use of oral supplements of vitamins and minerals are permitted although the current use of Vitamin A supplementation shall be documented.
* The site Principal Investigator may declare any patient at their site ineligible to participate in the study for a sound medical reason prior to the patient's enrollment into the study.
* Any systemic disease with a limited survival prognosis (e.g. cancer, severe/unstable cardiovascular disease).
* Any condition that would interfere with the patient attending their regular follow-up visits every 6 months for up to 24 months, e.g. personality disorder, use of major tranquilizers such as Haldol or Phenothiazine, chronic alcoholism, Alzheimer's Disease or drug abuse.
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular, neurological, pulmonary, renal, hepatic, endocrine or gastro-intestinal disorders.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population shall consist of up to 250 Stargardt disease patients (minimum of 150 patients) recruited at up to 14 clinical centers across the US and Europe. Must be at least 6 years old, able to cooperate in performing the examinations and be willing to attend regular 6 month follow-up visits for up to 24 months. Must present with atrophic lesions secondary to STGD and previously genotyped (at least 2 confirmed pathogenic mutations in the ABCA4 gene). If only 1 ABCA4 allele contains a pathogenic mutation, then the patient needs typical phenotype, i.e. at least one eye must have flecks at the level of the retinal pigment epithelium typical for STGD. Best-corrected visual acuity (BCVA) must be 20 ETDRS letters (20/400 Snellen equivalent) or better.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2013-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Scholl, MD, Study Chair — Wilmer Eye Institute at the Johns Hopkins University
Locations (9):
- United States (6):
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Wilmer Eye Institute, Johns Hopkins University, Baltimore, Maryland
  - Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
  - Moran Eye Center, University of Utah, Salt Lake City, Utah
- Institut de la Vision, Paris, France
- Center for Ophthalmic Research, University of Teubingen, Tübingen, Germany
- Moorfields Eye Hospital, London, United Kingdom

REFERENCES:
- [Background] Schonbach EM, Ibrahim MA, Strauss RW, Birch DG, Cideciyan AV, Hahn GA, Ho A, Kong X, Nasser F, Sunness JS, Zrenner E, Sadda SR, West SK, Scholl HPN; Progression of Stargardt Disease Study Group. Fixation Location and Stability Using the MP-1 Microperimeter in Stargardt Disease: ProgStar Report No. 3. Ophthalmol Retina. 2017 Jan-Feb;1(1):68-76. doi: 10.1016/j.oret.2016.08.009. Epub 2016 Oct 31. PMID 31047397
- [Background] Kong X, West SK, Strauss RW, Munoz B, Cideciyan AV, Michaelides M, Ho A, Ahmed M, Schonbach EM, Cheetham JK, Ervin AM, Scholl HPN; ProgStar study group. Progression of Visual Acuity and Fundus Autofluorescence in Recent-Onset Stargardt Disease: ProgStar Study Report #4. Ophthalmol Retina. 2017 Nov-Dec;1(6):514-523. doi: 10.1016/j.oret.2017.02.008. Epub 2017 Apr 28. PMID 31047445
- [Background] Strauss RW, Munoz B, Ho A, Jha A, Michaelides M, Mohand-Said S, Cideciyan AV, Birch D, Hariri AH, Nittala MG, Sadda S, Scholl HPN; ProgStar Study Group. Incidence of Atrophic Lesions in Stargardt Disease in the Progression of Atrophy Secondary to Stargardt Disease (ProgStar) Study: Report No. 5. JAMA Ophthalmol. 2017 Jul 1;135(7):687-695. doi: 10.1001/jamaophthalmol.2017.1121. PMID 28542697
- [Background] Schonbach EM, Wolfson Y, Strauss RW, Ibrahim MA, Kong X, Munoz B, Birch DG, Cideciyan AV, Hahn GA, Nittala M, Sunness JS, Sadda SR, West SK, Scholl HPN; ProgStar Study Group. Macular Sensitivity Measured With Microperimetry in Stargardt Disease in the Progression of Atrophy Secondary to Stargardt Disease (ProgStar) Study: Report No. 7. JAMA Ophthalmol. 2017 Jul 1;135(7):696-703. doi: 10.1001/jamaophthalmol.2017.1162. PMID 28542693
- [Result] Strauss RW, Ho A, Munoz B, Cideciyan AV, Sahel JA, Sunness JS, Birch DG, Bernstein PS, Michaelides M, Traboulsi EI, Zrenner E, Sadda S, Ervin AM, West S, Scholl HP; Progression of Stargardt Disease Study Group. The Natural History of the Progression of Atrophy Secondary to Stargardt Disease (ProgStar) Studies: Design and Baseline Characteristics: ProgStar Report No. 1. Ophthalmology. 2016 Apr;123(4):817-28. doi: 10.1016/j.ophtha.2015.12.009. Epub 2016 Jan 16. PMID 26786511
- [Result] Kong X, Strauss RW, Michaelides M, Cideciyan AV, Sahel JA, Munoz B, West S, Scholl HP; ProgStar Study Group. Visual Acuity Loss and Associated Risk Factors in the Retrospective Progression of Stargardt Disease Study (ProgStar Report No. 2). Ophthalmology. 2016 Sep;123(9):1887-97. doi: 10.1016/j.ophtha.2016.05.027. Epub 2016 Jul 2. PMID 27378015
- [Result] Kong X, Strauss RW, Cideciyan AV, Michaelides M, Sahel JA, Munoz B, Ahmed M, Ervin AM, West SK, Cheetham JK, Scholl HPN; ProgStar Study Group. Visual Acuity Change over 12 Months in the Prospective Progression of Atrophy Secondary to Stargardt Disease (ProgStar) Study: ProgStar Report Number 6. Ophthalmology. 2017 Nov;124(11):1640-1651. doi: 10.1016/j.ophtha.2017.04.026. Epub 2017 May 23. PMID 28549516
- [Result] Strauss RW, Munoz B, Ho A, Jha A, Michaelides M, Cideciyan AV, Audo I, Birch DG, Hariri AH, Nittala MG, Sadda S, West S, Scholl HPN; ProgStar Study Group. Progression of Stargardt Disease as Determined by Fundus Autofluorescence in the Retrospective Progression of Stargardt Disease Study (ProgStar Report No. 9). JAMA Ophthalmol. 2017 Nov 1;135(11):1232-1241. doi: 10.1001/jamaophthalmol.2017.4152. PMID 29049437
- [Result] Kong X, Fujinami K, Strauss RW, Munoz B, West SK, Cideciyan AV, Michaelides M, Ahmed M, Ervin AM, Schonbach E, Cheetham JK, Scholl HPN; ProgStar Study Group. Visual Acuity Change Over 24 Months and Its Association With Foveal Phenotype and Genotype in Individuals With Stargardt Disease: ProgStar Study Report No. 10. JAMA Ophthalmol. 2018 Aug 1;136(8):920-928. doi: 10.1001/jamaophthalmol.2018.2198. PMID 29902293
- See also: Study Website — http://progstar.org
- See also: Study Sponsor website — http://fightblindness.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Retrospective Cohort: Patients with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). Participant's data are from clinical examinations and central reading center (RC) grading of retinal imaging (fundus auto-fluorescence, and spectral domain optical coherence tomography (OCT).
- Prospective Cohort: Patients with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). Participant's data are from standardized clinical examinations and central reading center (RC) grading of retinal imaging (fundus auto-fluorescence, spectral domain optical coherence tomography (OCT) and micro-perimetry (optional).
Period: Total Study - Retrospective
Arm/Group | Retrospective Cohort | Prospective Cohort
Started | 251 | 0
Completed | 251 | 0
Not Completed | 0 | 0
Period: Total Study - Prospective
Arm/Group | Retrospective Cohort | Prospective Cohort
Started | 0 | 259
Completed | 0 | 230
Not Completed | 0 | 29
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 8
Not completed — Withdrawal by Subject | 0 | 13
Not completed — Not available at time of visit | 0 | 5
Not completed — No show | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: In Retrospective cohort, 251 participants contributed 433 eyes. In Prospecitive cohort, 259 participants contributed 489 eyes.
Groups:
- Retrospective Cohort: Subjects with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). Clinical data from multiple centers extracted from medical records. Participants were to have at least two visits with at least one of the study image modalities (fundus auto-fluorescence, micro-perimetry, or spectral domain optical coherence tomography (OCT))
- Prospective Cohort: Multicenter prospective longitudinal cohort. Patients with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). Participants were to have standardized visits at baseline and every 6 months for 24 months. Participant's data are from clinical examinations and central RC grading of retinal imaging (fundus auto-fluorescence, spectral domain optical coherence tomography (OCT)) and micro-perimetry.
- Total: Total of all reporting groups
Arm/Group | Retrospective Cohort | Prospective Cohort | Total
Number analyzed (Participants) | 251 | 259 | 510
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 69 | 51 | 120
  Between 18 and 65 years | 179 | 201 | 380
  >=65 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 141 | 290
  Male | 102 | 118 | 220
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Middle Eastern | 174 | 222 | 396
  Race: Black or African American | 14 | 20 | 34
  Race: Asian/Indian | 10 | 10 | 20
  Race: Other | 5 | 1 | 6
  Race: More than one race | 2 | 2 | 4
  Race: Don't know/missing | 46 | 4 | 50
Region of Enrollment [Number; unit: participants]
  United States | 90 | 137 | 227
  United Kingdom | 79 | 30 | 109
  France | 49 | 48 | 97
  Germany | 33 | 44 | 77

OUTCOME MEASURES:

1. Primary Outcome: Yearly Progression Rate of Atrophic Lesions Using Fundus Autofluorescence (FAF) Images
Description: Yearly increase in area of decreased auto-fluorescence (DAF) which is defined as the sum of definite and questionable decreased auto-fluorescence
Time Frame: 2-12 years
Population: Eyes of participants with at least 2 visits with gradable fundus auto-fluorescence images with atrophic lesions present
Measure: Mean (95% Confidence Interval); unit: mm^2/year
Units Other Than Participants: eyes
Arm/Group | Retrospective Cohort | Prospective Cohort
Number analyzed (Participants) | 215 | 259
Number analyzed (eyes) | 386 | 489
mm^2/year | 0.35 [0.28 to 0.43] | 0.64 [0.57 to 0.71]

2. Secondary Outcome: Yearly Rate of Loss of Retinal Sensitivity as Measured by Scotopic Microperimetry (MP)
Description: The yearly rate of change in retinal sensitivity. Sensitivity tested with a Nidek MP-1 machine using a modified Humphrey 10-2 grid. The sensitivity was the average sensitivity from a 68-points test pattern (Prospective cohort only)
Time Frame: 2 years
Population: Microperimetry data are available for only the Prospective cohort at centers with required equipment
Measure: Mean (95% Confidence Interval); unit: dB/year
Units Other Than Participants: eyes
Arm/Group | Retrospective Cohort | Prospective Cohort
Number analyzed (Participants) | 0 | 238
Number analyzed (eyes) | 0 | 449
dB/year |  | -0.76 [-0.87 to -0.66]

3. Secondary Outcome: Yearly Rate of Visual Acuity Loss
Description: Yearly change of visual acuity. Visual acuity measures of best-corrected or presenting VA extracted from medical record charts. Prospective cohort is best-corrected visual acuity using Early-Treatment Diabetic Retinopathy study methods
Time Frame: 2-12 years
Measure: Mean (95% Confidence Interval); unit: logMAR/year
Units Other Than Participants: eyes
Arm/Group | Retrospective Cohort | Prospective Cohort
Number analyzed (Participants) | 176 | 259
Number analyzed (eyes) | 332 | 489
logMAR/year | 0.030 [0.026 to 0.043] | 0.011 [0.004 to 0.018]

4. Secondary Outcome: Difference in the Rate of Retinal Sensitivity Change Per Year Between Photopic and Scotopic Micro-perimetry Testing
Description: Difference in the yearly rate of change in retinal sensitivity under photopic and scotopic conditions. Sensitivity tested with a Nidek MP-1. Scotopic sensitivity was obtained using a 40 points test pattern, and photopic sensitivity was obtained using a 68 points test pattern in a subset of Prospective cohort patients
Time Frame: 2 years
Population: Photopic microperimetry was obtained in a subset of patients, in a single designated study eye
Measure: Mean (95% Confidence Interval); unit: dB/year
Units Other Than Participants: eyes
Arm/Group | Retrospective Cohort | Prospective Cohort
Number analyzed (Participants) | 0 | 118
Number analyzed (eyes) | 0 | 118
dB/year |  | -0.78 [-1.16 to -0.41]

5. Secondary Outcome: Yearly Rate of Loss of Overall Retinal Thickness
Description: Yearly decrease of overall retinal thickness using spectral domain optical coherence tomography (SD-OCT) scans from a 20° x 20° scan area centered on the fovea. Data are only available for the Prospective cohort.
Time Frame: Participants followed at Baseline, 6 months, 12 months and 24 months
Population: All visits of eligible eyes of the 258 participants with gradable overall thickness. Only OCT scans with adequate and fair quality are included
Measure: Mean (95% Confidence Interval); unit: microns/year
Units Other Than Participants: eyes
Groups:
- Prospective Cohort: Multicenter prospective longitudinal cohort. Patients with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). OCT scans were graded by a central reading center.
Arm/Group | Prospective Cohort
Number analyzed (Participants) | 258
Number analyzed (eyes) | 487
microns/year | -2.85 [-3.19 to -2.52]

6. Secondary Outcome: Yearly Rate of Loss of Outer Ring Retinal Thickness
Description: Yearly decrease of outer ring retinal thickness using SD-OCT scans from a 20° x 20° scan area centered on the fovea. Outer ring defined as ETDRS fields 1-4.
Time Frame: Participants followed at Baseline, 6 months, 12 months and 24 months
Population: All visits of eligible eyes of the 258 participants with gradable thickness in the outer ring. Only OCT scans with adequate and fair quality are included
Measure: Mean (95% Confidence Interval); unit: microns/year
Units Other Than Participants: eyes
Arm/Group | Prospective Cohort
Number analyzed (Participants) | 258
Number analyzed (eyes) | 487
microns/year | -2.84 [-3.19 to -2.50]

7. Secondary Outcome: Yearly Rate of Loss of the Inner Ring Retinal Thickness
Description: Yearly decrease of the inner ring retinal thickness using SD-OCT scans from a 20° x 20° scan area centered on the fovea. Inner ring defined as ETDRS fields 5-8. Data are only available for the Prospective cohort.
Time Frame: Participants followed at Baseline, 6 months, 12 months and 24 months
Population: All visits of eligible eyes of the 258 participants with gradable thickness in the inner ring. Only OCT scans with adequate and fair quality are included
Measure: Mean (95% Confidence Interval); unit: microns/year
Units Other Than Participants: eyes
Arm/Group | Prospective Cohort
Number analyzed (Participants) | 258
Number analyzed (eyes) | 487
microns/year | -3.20 [-3.68 to -2.72]

8. Secondary Outcome: Yearly Rate of Loss of the Central Ring Retinal Thickness
Description: Yearly decrease of the central ring retinal thickness using SD-OCT scans from a 20° x 20° scan area centered on the fovea. Central area defined as ETDRS fields 9. Data are only available for the Prospective cohort.
Time Frame: Participants followed at Baseline, 6 months, 12 months and 24 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: microns/year
Units Other Than Participants: eyes
Arm/Group | Prospective Cohort
Number analyzed (Participants) | 258
Number analyzed (eyes) | 487
microns/year | -2.24 [-3.06 to -1.42]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected in this natural history study
Description: As there was no intervention in this study, adverse events were not collected
Groups:
- Retrospective Cohort: Subjects with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). Clinical data from multiple centers extracted from medical records. Participants should had at least two visits with at least one of the study image modalities (fundus auto-fluorescence, micro-perimetry, or spectral domain optical coherence tomography (OCT)). Adverse events were not collected
- Prospective Cohort: Multicenter prospective longitudinal cohort. Patients with at least two pathogenic mutations in the ABCA4 gene (or one mutation, but the clinical phenotype of flecks at the level of the RPE typical for STGD1). Participants had standardized visits at baseline and every 6 months for 24 months. Participant's data are from clinical examinations and central RC grading of retinal imaging (fundus auto-fluorescence, spectral domain optical coherence tomography (OCT)) and micro-perimetry. Adverse events were not collected
Arm/Group | Retrospective Cohort | Prospective Cohort
All-Cause Mortality (participants affected / at risk) | 0/251 | 1/259
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-03-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT01977846/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT01977846/SAP_001.pdf